CLINICAL TRIAL: NCT04650763
Title: Effect of PRP on Bone Healing in Immediate Implants Analyzed by CBCT
Brief Title: Bone Healing in Immediate Dental Implants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CMH Lahore Medical College and Institute of Dentistry (Other)
Responsible Party: Principal Investigator, Prof. Abdul Mueed Zaigham, Professor & Head Prosthodontics Department, CMH Lahore Medical College and Institute of Dentistry
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Case # 466/ERC/CMH/LMC
Record Dates: First submitted 2020-11-14; First posted 2020-12-03 (Actual); Last update posted 2020-12-03 (Actual); Status verified 2020-11

CONDITIONS: Alveolar Bone Loss; Platelet Rich Plasma
Keywords: Dental implant, Cone Beam Computerized Tomography (CBCT).
MeSH Terms: conditions — Alveolar Bone Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Control Group (No Intervention): Dental implant was placed in these patients following full protocol of immediate implant placement.
- PRP Group (Experimental): In this group Platelet Rich Plasma (PRP) was injected in soft tissue over surgical site.
  Interventions: Biological: PRP injection; Device: Automated blood cell separator to extract PRP

INTERVENTIONS:
Biological: PRP injection — PRP was prepared using patient's blood and mixed with saline or mixture of calcium chloride and thrombin to form a liquid solution; in order to inject at the surgical site after placement of implant.
  Other Names: Platelet Rich Plasma injection
  Arms: PRP Group
Device: Automated blood cell separator to extract PRP — Blood was withdrawn from antecubital vein and mixed with anticoagulant. Blood sample was then centrifuged to obtain platelet rich plasma which was injected at surgical site after implant placement.
  Other Names: Automated blood cell separator/ centrifuge
  Arms: PRP Group

SUMMARY:
To study the effect of platelet-rich plasma concentrate on marginal bone loss and bone mineral density in immediate implant placement through CBCT.

DETAILED DESCRIPTION:
12 subjects were equally categorized into two groups. Group, I was the control group; whereas, the subjects in Group II received Platelet Rich Plasma (PRP) therapy. All subjects were given a standard treatment with single implant system. Inserted implants were analyzed through Cone Beam Computerized Tomography (CBCT). Records were registered at the baseline, at 12th week before functional loading and 26th week after functional loading.

ELIGIBILITY:
Inclusion Criteria:

* patients maintaining good oral hygiene, having adequate bone quantity at the implant site, uneventful extraction

Exclusion Criteria:

* Active infection around implant site, immunocompromised state, with current major systemic disease (uncontrolled diabetes, rheumatoid arthritis, etc.) or oral pathologies, history of bleeding disorders or on anticoagulant therapy, or patients on bisphosphonates were excluded from the study

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2017-10-02 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2018-03-30 (Actual)

PRIMARY OUTCOMES:
Measurement of bone loss at baseline (12 weeks) and later at 26weeks | Baseline -before functional loading at 12 weeks & at 26 weeks- after functional loading to assess changes in marginal bone loss in sagittal view using CBCT
  Measurement at mesial in mm

SECONDARY OUTCOMES:
Measurement of bone loss at baseline (12 weeks) and later at 26weeks | Baseline -before functional loading at 12 weeks & at 26 weeks- after functional loading to assess changes in marginal bone loss in sagittal view using CBCT
  Measurement at distal in mm

OTHER OUTCOMES:
Bone Mineral Density | Baseline -before functional loading at 12 weeks & at 26 weeks- after functional loading to assess changes in marginal bone loss in sagittal view using CBCT
  Measurement in Hounsfield number

CONTACTS AND LOCATIONS:
Overall Officials: Aleshba Saba khan, BDS; FCPS, Principal Investigator — Institute of Dentistry; CMH Lahore Medical College; Naauman Zaheer, BDS; PhD, Principal Investigator — Institute of Dentistry; CMH Lahore Medical College; Abdul Mueed Zaigham, BDS; FCPS, Study Chair — Institute of Dentistry; CMH Lahore Medical College; Maliha Shahbaz, BDS; MPhil, Study Director — Oral Biology Department; Rashid Latif Dental College, Lahore; Usman Zaheer, BDS; FCPS, Principal Investigator — Lahore Medical & Dental College
Locations (1):
- Institute of Dentistry; CMH Lahore Medical College, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Boora P, Rathee M, Bhoria M. Effect of Platelet Rich Fibrin (PRF) on Peri-implant Soft Tissue and Crestal Bone in One-Stage Implant Placement: A Randomized Controlled Trial. J Clin Diagn Res. 2015 Apr;9(4):ZC18-21. doi: 10.7860/JCDR/2015/12636.5788. Epub 2015 Apr 1. PMID 26023636
- [Derived] Khan AS, Zaheer N, Zaigham AM, Shahbaz M, Zaheer U, Alam MK. Effect of Platelet-Rich Plasma on Bone Healing in Immediate Implants Analyzed by Cone Beam Computerized Tomography: A Randomized Controlled Trial. Biomed Res Int. 2021 Mar 13;2021:6685991. doi: 10.1155/2021/6685991. eCollection 2021. PMID 33791377